CLINICAL TRIAL: NCT03687476
Title: An Open-label, Multicenter Safety and Tolerability Study of VTS-270 (2-hydroxypropyl-β-cyclodextrin) in Pediatric Subjects Aged < 4 Years With Neurologic Manifestations of Niemann-Pick Type C (NPC) Disease
Brief Title: Safety and Tolerability Study of VTS-270 in Pediatric Participants With Niemann-Pick Type C (NPC) Disease
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: Business decision to Cancel
Sponsor: Vtesse, LLC, a Mallinckrodt Pharmaceuticals Company (Industry)
Responsible Party: Sponsor
Organization: Mallinckrodt (Industry)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VTS270-303
Record Dates: First submitted 2018-08-06; First posted 2018-09-27 (Actual); Last update posted 2020-07-22 (Actual); Status verified 2020-07

CONDITIONS: Niemann-Pick Disease, Type C
MeSH Terms: conditions — Niemann-Pick Disease, Type C

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VTS-270 (Part A) (Experimental): VTS-270 200 milligram per milliliter (mg/mL) will be administered intrathecally by lumbar puncture every 2 weeks followed by dose escalation of 100 mg/mL increments up to a maximum tolerable dose of 900 mg/mL. The highest tolerable dose is considered as clinically relevant dose which will be administered throughout the remaining duration of the 20-week treatment period of Part A.
  Interventions: Drug: VTS-270
- VTS-270 (Part B) (Experimental): VTS-270 200 mg/mL will be administered intrathecally by lumbar puncture every 2 weeks in Part B followed by a re-challenge to dose escalation of 100 mg/mL increments up to a maximum tolerable dose of 900 mg/mL. In case of intolerance, the dose should be returned to previously tolerable dose and should be continued throughout the duration of Part B (end of study).
  Interventions: Drug: VTS-270

INTERVENTIONS:
Drug: VTS-270 — VTS-270 200 mg/mL administered as described in the arm group description.

SUMMARY:
This is a Phase-2, multicenter, multiple dose, open-label, 2-part evaluation study which will primarily assess the safety and tolerability of VTS-270 (2-hydroxypropyl beta-cyclodextrin [HP-β-CD]) in pediatric participants with age <4 years.

DETAILED DESCRIPTION:
In Part A of the study, participants after confirmation of the diagnosis of NPC will receive VTS-270 for 20 weeks during the active treatment period. Further, based on investigator's discretion participants would either end treatment with a follow-up visit 28 days (+/- 7) days after last treatment, or will enter to Part-B to benefit from open-label treatment.

ELIGIBILITY:
Inclusion Criteria:

1. The parent(s)/legal guardian(s) must be adequately informed and understand the nature and risks of the study. The participant's parent or legal guardian must provide a signature and date on the informed consent form (ICF).
2. Participants must have neurologial symptoms defined as, any area of developmental delay 1 SD below the mean (example, developmental quotient or standard score under 85 in any domain on the Mullen Scale Early Learning [MSEL]) or a significant developmental quotient /standard score drop on the MSEL.
3. Diagnosis of NPC determined by one of the following:

   1. Two NPC1 or NPC2 mutations;
   2. Positive filipin staining or oxysterol testing and at least one NPC1 or NPC2 mutation;
   3. Vertical supranuclear gaze palsy in combination with either:

   i. One NPC1/NPC2 mutation, or

   ii. Positive filipin staining or oxysterol levels consistent with NPC1 or NPC2 disease.
4. If taking miglustat (Zavesca), participant(s) must have been on a stable dose for 6 weeks prior to the Screening Visit and willing to remain on a stable dose for the duration of participation in this study. If not taking migulstat, the participant must have been off treatment for a minimum of 6 weeks prior to the Baseline Visit.
5. If a participant has a history of seizures, the condition must be adequately controlled (the pattern of seizure activity must be stable) and the participant must be on a stable dose and regimen of antiepileptic medication(s) 4 weeks prior to the Screening Visit.
6. Prior exposure to VTS-270 is permitted.
7. The participant's parent(s)/legal guardian(s) are able to communicate effectively with study personnel.
8. Parent(s)/legal guardian(s) are able and willing to follow all protocol requirements and study restrictions.
9. Parent(s)/legal guardian(s) are able and willing to return participants for all study visits.

Exclusion Criteria:

1. Is from a vulnerable population, as defined by the US CFR Title 45, Part 46, Section 46.111(b) and other local and national regulations, including but not limited to, employees (temporary, part-time, full time, etc) or a family member of the research staff conducting the study, or of the sponsor, or of the contract research organization, or of the institutional review board (IRB)/independent ethics committee (IEC).
2. Has a history of sensitivity or allergy to any product containing HP-β-CD.
3. A history of hypersensitivity reactions or allergy to the anesthetic and/or sedative agents to be used for the lumbar puncture procedure.
4. Taken an anticoagulant in the 2 weeks prior to the Baseline Visit or plan to use anticoagulants during the study.
5. Change in antiepileptic treatment between the Screening Visit and the Baseline Visit.
6. Received treatment for any investigational product (exclusive of VTS-270) within 4 weeks of the Baseline Visit or at least 5 half-lives, whichever criteria is longest.
7. A suspected infection of the central nervous system or any systemic infection.
8. A spinal deformity that is likely to impact the ability to perform repeated LPs.
9. Evidence of obstructive hydrocephalus or normal pressure hydrocephalus.
10. Undergoing intravenous treatment with VTS-270. Note: prior or current treatment with IT VTS-270 is not exclusionary.
11. A known bleeding disorder.
12. Has any of the following laboratory abnormalities ( greater than 1.5 times the upper limit of normal) at the Screening Visit:

    * Neutropenia
    * Thrombocytopenia
    * Activated partial thromboplastin time
    * Prothrombin time prolongation.
13. Has any other clinically significant disease, disorder or laboratory abnormality, which, in the opinion of the investigator, might put the participant at risk due to participation in the study, or may influence the results of the study or the participant's ability to complete the study.
14. Is participating in or plans to participate in any other interventional research study from the time of screening and throughout this study.
15. Also excluded are participant, who in the opinion of the investigator, are unable to comply with the protocol or who have a medical condition (eg, cardiovascular, respiratory, hematologic, neurologic, psychiatric, renal) that would potentially increase the risk of study participation.

Max Age: 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2020-05 (Estimated); Primary Completion 2022-10-30 (Estimated); Study Completion 2022-10-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Part A | Baseline up to Week 20 (End of Part A)
  An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. SAEs were AEs excluding non-serious AEs.
Number of Participants With Clinically Significant Vital Signs: Part A | Baseline up to Week 20 (End of Part A)
  Clinically significant vital sign is defined as an abnormal vital sign result that results in a treatment-emergent AEs. Abnormal clinically significant vital signs included absolute systolic blood pressure (BP) values less than (<) 90 millimeter of mercury (mmHg), maximum increase or decrease of greater than or equal to (>=) 30 mmHg from baseline for systolic BP; absolute diastolic BP <50 mmHg with maximum increase or decrease of >=20 mmHg from baseline and absolute heart rate values <40 beats per minute (bpm), >120 bpm for supine or sitting measurement, >140 bpm for standing measurement, temperature <32 or >40 degree centigrade, respiratory rate of <10 or >50 breaths/minute.
Number of Participants With Clinically Significant Change from Baseline in Body Weight: Part A | Baseline up to Week 20 (End of Part A)
  Any change from baseline in body weight is considered by the investigator to be clinically significant and will be recorded as treatment-emergent AE.
Number of Participants With Clinically Significant Change from Baseline in Body Height: Part A | Baseline up to Week 20 (End of Part A)
  Any change from baseline in body height is considered by the investigator to be clinically significant and will be recorded as treatment-emergent AE.
Number of Participants With Clinically Significant Laboratory Test Abnormalities: Part A | Baseline up to Week 20 (End of Part A)
  Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (< 0.8*lower limit of normal[LLN]); leucocytes (<0.6/>1.5*upper limit of normal [ULN]); platelets (<0.5*LLN/>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN/>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN/>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN/>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN/>1.1*ULN); urine red blood cells (RBCs), urine white blood cells (WBCs), urine epithelial cells (>=6 high-powered field), urine bacteria >20 high-powered field; qualitative urine glucose, ketones, protein values >=1 in urine dipstick test. Total number of participants with any laboratory abnormalities was reported.

SECONDARY OUTCOMES:
Number of Participants With Treatment-Emergent Adverse Events (AEs) or Serious Adverse Events (SAEs): Part B | Week 22 up to 3 years (End of Study or Part B)
  An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent are events between first dose of study drug and up to 28 days after last dose that were absent before treatment or that worsened relative to pre-treatment state. SAEs were AEs excluding non-serious AEs.
Number of Participants With Clinically Significant Vital Signs: Part B | Week 22 up to 3 years (End of Study or Part B)
  Clinically significant vital sign is defined as an abnormal vital sign result that results in a treatment-emergent AEs. Abnormal clinically significant vital signs included absolute systolic blood pressure (BP) values less than (<) 90 millimeter of mercury (mmHg), maximum increase or decrease of greater than or equal to (>=) 30 mmHg from baseline for systolic BP; absolute diastolic BP <50 mmHg with maximum increase or decrease of >=20 mmHg from baseline and absolute heart rate values <40 beats per minute (bpm), >120 bpm for supine or sitting measurement, >140 bpm for standing measurement, temperature <32 or >40 degree centigrade, respiratory rate of <10 or >50 breaths/minute.
Number of Participants With Clinically Significant Change from Baseline in Body Weight: Part B | Week 22 up to 3 years (End of Study or Part B)
  Any change from baseline in body weight is considered by the investigator to be clinically significant and will be recorded as treatment-emergent AE.
Number of Participants With Clinically Significant Change from Baseline in Body Height: Part B | Week 22 up to 3 years (End of Study or Part B)
  Any change from baseline in body height is considered by the investigator to be clinically significant and will be recorded as treatment-emergent AE.
Number of Participants With Clinically Significant Laboratory Test Abnormalities: Part B | Week 22 up to 3 years (End of Study or Part B)
  Criteria for laboratory tests abnormalities included: hemoglobin, hematocrit and red blood cells (< 0.8*lower limit of normal[LLN]); leucocytes (<0.6/>1.5*upper limit of normal [ULN]); platelets (<0.5*LLN/>1.75*ULN); neutrophils, lymphocytes (<0.8*LLN/>1.2*ULN); eosinophils, basophils, monocytes (>1.2*ULN); total bilirubin (>1.5*ULN); aspartate aminotransferase (AST), alanine aminotransferase (ALT), alkaline phosphatase (>3*ULN), total protein, albumin (<0.8*LLN/>1.2*ULN); creatinine, urea (>1.3*ULN); glucose (<0.6*LLN/>1.5*ULN); uric acid (>1.2*ULN); sodium, potassium, chloride, calcium, bicarbonate (<0.9*LLN/>1.1*ULN); urine red blood cells (RBCs), urine white blood cells (WBCs), urine epithelial cells (>=6 high-powered field), urine bacteria >20 high-powered field; qualitative urine glucose, ketones, protein values >=1 in urine dipstick test. Total number of participants with any laboratory abnormalities was reported.
Change From Baseline in Audiological Examinations at Week 6, 12, 20, 44, and every 24 Week Thereafter Until End of Treatment (EOT: 3 Years) | Baseline, Week 6, 12, 20, 44, every 24 Week thereafter until EOT (3 years)
  Standard developmentally appropriate audiological examinations suited to the individual participants will be used to assess auditory system function (physical tests: tympanometry and otoacoustic emissions) and hearing sensitivity (behavioral test: word recognition and pure-tone and speech thresholds).
Change From Baseline in Cognitive and Motor Development Assessed Using Mullen Scale of Early Learning (MSEL) at Week 6, 12, 20, 44, and every 24 Week Thereafter Until End of Treatment (EOT: 3 Years) | Baseline, Week 6, 12, 20, 44, every 24 Week thereafter until EOT (3 years)
  The MSEL is a standardized developmental test for children consisting of five subscales: fine motor, visual reception, expressive language, receptive language and an optional fifth gross motor scale (scale includes standing, walking and running) that only measures skills to 36 months. The raw score is reported for each subscale domain. The potential score ranges are as follows: Visual Reception: 33 items, score range=0-50, Fine Motor: 30 items, score range= 0-49, Receptive Language: 33 items, score range= 0-48, Expressive Language: 28 items, score range= 0-50. A higher raw score indicates more advanced abilities in that section.
Change From Baseline in Auditory Brainstem Response (ABR) Assessed Using Standard Clinical Pediatric Score at Week 6, 12, 20, 44, and every 24 Week Thereafter Until End of Treatment (EOT: 3 Years) | Baseline, Week 6, 12, 20, 44, every 24 Week thereafter until EOT (3 years)
  The ABR is a voltage response evoked by acoustic stimuli as sound is processed along the auditory pathway. It consists of electrical signals resulting from the sum of sound-evoked activity along the auditory nerve and brainstem nuclei. The ABR analysis determines the sound intensity at which a neural response first appears (hearing threshold). Other parameters of interest include amplitude (the number of neurons firing), latency (the speed of transmission), interpeak latency (the time between peaks), and interaural latency (the difference in wave V latency between ears). The interpeak latency I-V interval (or central transmission time) is considered the most reliable index of brainstem function. Auditory brainstem response assessments were based on standard clinical pediatric score criteria: mild hearing loss: 21-40 decibels hearing level (dBHL), moderate hearing loss: 41-70 dBHL, severe hearing loss: 71-90 dBHL, profound hearing loss: 91dBHL.
Change From Baseline in Clinician Global Impression of Change (CGIC) Using Likert Score at Week 6, 12, 20, 44, and every 24 Week Thereafter Until End of Treatment (EOT: 3 Years) | Baseline, Week 6, 12, 20, 44, every 24 Week thereafter until EOT (3 years)
  The Clinician-CGIC is conducted by a clinician who is trained in performing neurological examinations. CGIC is measured using 7-point Likert scale ranging from 1 = "very much improved" to 7 = "very much worse". If the rater notes an improvement or worsening on the scale, the rater should indicate the major factor for the reported changes in score.
Change From Baseline in Caregiver Global Impression of Change (CGIC) Using Likert Score at Week 6, 12, 20, 44, and every 24 Week Thereafter Until End of Treatment (EOT: 3 Years) | Baseline, Week 6, 12, 20, 44, every 24 Week thereafter until EOT (3 years)
  The caregiver-CGIC is to be completed by the responsible parent or legal guardian. CGIC is measured using 7-point Likert scale ranging from 1 = "very much improved" to 7 = "very much worse". If the caregiver notes an improvement or worsening on the scale, the caregiver should indicate the major reason for the reported changes in score.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Mallinckrodt

IPD SHARING:
Plan to Share IPD: No